CLINICAL TRIAL: NCT05112471
Title: Efficacy of Combined Air-abrasive+Ultrasonic (Guided Biofilm Therapy GBT) vs. Standard Root Debridement (Scaling and Root Planing+ Ultrasonic SRP+US) in the Treatment of Severe Generalized Periodontitis: A Randomized Clinical Trial
Brief Title: Efficacy of GBT vs SRP+US, in the Treatment of Severe Generalized Periodontitis.
Acronym: ERISRP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Principal Investigator, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ERISRP
Record Dates: First submitted 2021-10-21; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Periodontitis, Aggressive; Periodontal Diseases; Periodontitis
Keywords: Periodontitis; Biofilm; Air-polishing; SRP; Ultrasonic
MeSH Terms: conditions — Aggressive Periodontitis; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Intervention Model Description: Split Mouth, RCT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided Biofilm Therapy (Experimental): Airflow with erythritol powder to remove supra and sub gingival biofilm and plaque, perioflow with erythritol powder at deep pathological pockets (PPD > 4mm) and ultrasonic debridement with an ultrasonic scaler for remove supra and sub gingival calculus.
  Interventions: Device: Airflow, Perioflow and Erythritol powder and ultrasonic debridement
- Scaling and Root Planning - Ultrasonic Debridement (Active Comparator): Ultrasonic debridement with an ultrasonic scaler for remove supra and sub gingival calculus, manual debridement with curettes at deep pathological pockets (PPD > 4mm) and rubber cup with polishing to remove supra gingival biofilm and plaque.
  Interventions: Device: Ultrasonic debridement and curettes

INTERVENTIONS:
Device: Airflow, Perioflow and Erythritol powder and ultrasonic debridement — Airflow and Perioflow combined with Erythritol powder will be used as an adjunct therapy
  Arms: Guided Biofilm Therapy
Device: Ultrasonic debridement and curettes — traditional Scaling and Root Planing with curettes and ultrasonic scaler
  Arms: Scaling and Root Planning - Ultrasonic Debridement

SUMMARY:
The first step in the management of periodontal disease involves the non-surgical removal of the soft and hard bacterial deposits at all supra- and sub-gingival sites, especially into deep pockets, which can be carried on with different instruments.

Unfortunately it seems that, after the initial therapy, many patients still present with active pockets (residual pockets) requiring further treatment and posing a risk of disease progression. This might be due to limitations of the instruments applied and patient-related factors. Air-polishing with low-abrasiveness powders seems to be very effective in the removal of supra- and sub-gingival biofilm and could provide additional benefits during the treatment of pockets.

The aim of this randomized, controlled, split-mouth study was to compare the efficacy of full-mouth air-polishing followed by ultrasonic debridement (GBT) versus traditional Scaling and Root Planing (SRP), in terms of pocket closure in patients with stage III-IV periodontitis.

To test this hypothesis, the mouth of each patients, upon initial evaluation, were divided in 2 parts:

1. The control group undergoing a standard procedure: ultrasonic debridement with an ultrasonic scaler for remove supra and sub gingival calculus, manual debridement with curettes at deep pathological pockets (PPD > 4mm) and rubber cup with polishing to remove supra gingival biofilm and plaque.
2. The study group undergoing the innovative air polishing procedure: airflow with erythritol powder to remove supra and sub gingival biofilm and plaque, perioflow at deep pathological pockets (PPD > 4mm) and ultrasonic debridement with an ultrasonic scaler for remove supra and sub gingival calculus.

The prevalence of residual pockets will be evaluated at 6 weeks and 3 months after the initial therapy and compared between the two groups.

DETAILED DESCRIPTION:
TRIAL DESIGN:

A prospective, single-masked, randomized, split-mouth, longitudinal clinical trial.

OUTCOME:

1. The primary outcome was the number of experimental sites (PPD >4mm and <10mm) becoming closed pockets (PPD ≤ 4mm) at 6 weeks (T1) and 3 months (T2) after initial therapy.
2. Secondary outcomes were the variations in PPD, REC (Clinical Gingival Recession), CAL (Clinical Attachment Level), BOP (Bleeding On Probing) and PI (Plaque Index) at the experimental sites and treatment time.

A 10% difference in the primary outcome between the two protocols was set as the threshold to define inferiority/non-inferiority of the Test treatment.

STUDY POPULATION:

thirty-two (32) adults, aged 18-75 years, will be entered into study (randomized).

Randomized subjects who deviate from the protocol (major protocol deviation) and, for this reason, are excluded from the analysis, will be replaced to guarantee that the sample required for the analysis (32) is reached.

INCLUSION CRITERIA:

* Signed Informed Consent Form.
* Male and female subjects, aged 18-75 years, inclusive.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* Diagnosis of Stage III-IV periodontitis;17
* At least 6 sites per quadrant with Pocket Probing Depth (PPD) ≥ 3mm;
* At least 5 teeth per quadrant;
* Availability for the 3-month duration of the study for an assigned subject.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form.
* Male and female subjects, aged 18-75 years, with diagnosis of severe generalized periodontitis.
* Good general health (free of systemic diseases such as diabetes, HIV infection or genetic disorder, ongoing malignant disease of any type that could influence the outcome of the treatment and might interfere with the evaluation of the study objectives).
* Diagnosis of Stage III-IV periodontitis;
* At least 6 sites per quadrant with Pocket Probing Depth (PPD) ≥ 3mm;
* At least 5 teeth per quadrant;
* Availability for the 3-month duration of the study for an assigned subject.

Exclusion Criteria:

* Severe Smoking more than 10 cigarettes per day
* Pregnancy or nursing.
* Radiotherapy or Chemotherapy.
* BPCO (chronic obstructive pulmonary disease), asma.
* Systemic long-term corticosteroid treatment.
* Antibiotic treatment in the period of 3 months before the start of the study.
* Non surgical therapy in the period of 3 months before the start of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-11-22 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2020-04-04 (Actual)

PRIMARY OUTCOMES:
The number of experimental sites (PPD > 4mm and <10mm) becoming closed pockets (PPD ≤ 4mm). | 3 months after initial therapy.
  A 10% difference in the primary outcome between the two protocols was set as the threshold to define inferiority/non-inferiority of the Test treatment.

SECONDARY OUTCOMES:
Change in PPD (periodontal depth) | 3 months after initial therapy.
  Change in mean PD value for each patient measured (from the gingival margin to the bottom of the pocket). Baseline values will be compared to the values recorded in the follow-up visits.
Change in REC (Clinical Gingival Recession) | 3 months after initial therapy.
  Change in mean of REC value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Change in CAL (Clinical Attachment Level) | 3 months after initial therapy.
  Change in mean of CAL value for each patient should be calculated. Baseline values will be compared to the values recorded in the follow-up visits.
Change in BOP (Bleeding on Probing) | 3 months after initial therapy.
  Change in percentage of sites positive to bleeding on probing. Baseline values will be compared to the values recorded in the follow-up visits.
Change in PI (Plaque Index) | 3 months after initial therapy.
  Change in percentage of site with plaque. Baseline values will be compared to the values recorded in the follow-up visits.

CONTACTS AND LOCATIONS:
Overall Officials: Magda Mensi, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- Magda Mensi, Brescia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-16): https://cdn.clinicaltrials.gov/large-docs/71/NCT05112471/Prot_SAP_000.pdf